CLINICAL TRIAL: NCT01559870
Title: Peri-operative Prediction of Prolonged Stay in the Cardiac Intensive Care Unit for Adult Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Peri-operative Prediction of Prolonged Stay in the Cardiac Intensive Care Unit for Adult Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Thepakorn Sathitkarnmanee (Other)
Collaborators: Khon Kaen University (Other)
Responsible Party: Sponsor-Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Organization: Khon Kaen University (Other)
Other Study IDs: HE541122
Record Dates: First submitted 2012-03-13; First posted 2012-03-21 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-03

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery; Cytokine Release Syndrome
Keywords: cardiac surgery; cytokine; clinical scoring system; risk factor
MeSH Terms: conditions — Cytokine Release Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood taken from arterial line
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with elective cardiac surgery: adult patients who had undergone elective cardiac surgery with CPB

SUMMARY:
The purpose of this study is to create a model using intra-operative modified SOFA score and peri-operative clinical factors to predict prolonged stay in the cardiac intensive care unit (CICU) for adult cardiac surgery with heart-lung machine

DETAILED DESCRIPTION:
Cardiac surgery using cardiopulmonary bypass (CPB) is commonly associated with a systemic inflammatory response that exacerbates peri-operative life-threatening complications and multiple organ dysfunction syndromes. These features can prolong the stay in the CICU. Many peri-operative clinical risk factors contribute to those adverse outcomes resulting in prolonged CICU stay. If the investigators can create a model to identify the effects of these intra-operative clinical risk factors to prolonged CICU stay

ELIGIBILITY:
Inclusion Criteria:

* adult patients who had undergone elective cardiac surgery with CPB

Exclusion Criteria:

* under 18 years of age
* needing emergency surgery
* needing intra-aortic balloon pump

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who had undergone elective cardiac surgery with CPB
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Adjusted odds ratio of peri-operative clinical risk factors in prolonged CICU patients | 24 hours after CPB
  Blood samples were collected for cytokines investigation and leukocyte counts. Clinical scoring systems , major peri-operative clinical risk factors were calculated and recorded at each time point. Univariate odds ratio were calculated for each factors for prolonged CICU stay. Those significant factors were included in logistic regression model for analysis of adjusted odds ratios. Then, a model for prolonged CICU stay is constructed.

CONTACTS AND LOCATIONS:
Locations (3):
- Thailand (3):
  - Queen Sirikit Heart Cenrter, Khon Kaen, Changwat Khon Kaen
  - Queen Sirikit Heart Center, Khon Kaen, Changwat Khon Kaen
  - Queen Sirikit Heart Center, Khon Kaen